CLINICAL TRIAL: NCT05471674
Title: Neoadjuvant Immunotherapy With Anti-PD1 in Borderline Resectable Hepatocellular Carcinoma
Brief Title: Neoadjuvant Anti-PD1 in HCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr Tan-to CHEUNG (Other)
Responsible Party: Sponsor-Investigator, Dr Tan-to CHEUNG, Clinical Associate Professor, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-7KU
Record Dates: First submitted 2022-07-04; First posted 2022-07-25 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Hepatocellular Carcinoma; HCC; Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Nivolumab; Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Nivolumab; Procedure: Hepatectomy

INTERVENTIONS:
Drug: Nivolumab — 3 mg/kg on Day 1 of each 2-weekly cycle for 3 doses
Procedure: Hepatectomy — Hepatectomy will be performed approximately 2 weeks after the 3rd dose of nivolumab

SUMMARY:
This is a phase 2, single-arm trial designed to assess the clinical benefit of treatment with nivolumab administered in patients with untreated, borderline resectable HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent form prior to the screening procedures.
2. Age ≥ 18 years.
3. Histological proof of HCC.
4. Willingness to undergo a pre-dosing fresh tumour biopsy. Patients for whom fresh biopsy may not be feasible will be ineligible for enrollment.
5. Intermediate or locally-advanced HCC (according to HKLC tumour status categorization) with the option of resection for potential cure as assessed by surgeon.
6. Child-Pugh score ≤ 7 with no symptomatic ascites or ascites requiring therapeutic paracentesis.
7. ECOG performance status ≤ 1.
8. Life expectancy of ≥ 12 weeks.
9. Adequate organ function (blood transfusion or use of biologic response modifiers is not permitted).
10. Measurable disease according to RECIST v1.1.
11. Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception.
12. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception.
13. Able and willing to meet all protocol-required treatments, investigations and visits.

Exclusion Criteria:

1. Patients who have history of organ transplantation.
2. History of allergy or hypersensitivity to study drug components.
3. Patients who have active, known or suspected autoimmune disease. Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition adequately treated with hormonal replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger or deemed by the investigator not to affect safety assessment.
4. Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days prior to start of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
5. Patients who have received prior therapy with an anti-PD-1, anti-PD-L1, anti-PDL-2, or anti-CTLA-4 antibody (or any other antibody targeting T cell co-regulatory pathways).
6. Receipt of any cancer therapy in the pre-operative period.
7. Treatment with botanical preparations (e.g., herbal supplements or traditional Chinese medicine) intended for general health support or to treat the disease under study within 2 weeks prior to treatment.
8. Active, acute, or chronic clinically significant infections requiring therapy with the exception of hepatitis B or C virus infection. Patients with chronic HBV infection must be on antiviral therapy and have HBV DNA < 500 IU/ml. Active or chronic co-infection with hepatitis B and C, or hepatitis B and D is not allowed.
9. Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
10. Symptomatic congestive heart failure, defined as ≥ Class II of the New York Heart Association functional classification system or known LVEF < 50% at baseline.
11. Active angina pectoris or recent myocardial infarction (within 6 months).
12. Chronic atrial fibrillation or QTcF > 470 msec.
13. History of other previous cancer that would interfere with the determination of safety or efficacy of nivolumab with respect to HCC.
14. Women who are pregnant or breast-feeding.
15. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Pathological tumour response rate | After surgery (normally 6 weeks after the start of nivolumab)
  Proportion of patients with resected tumours having ≥30% necrosis

SECONDARY OUTCOMES:
Recurrence-free survival | At least 3 months after surgery
  The time from resection to disease recurrence or death from any cause
Overall survival | At least 3 months after surgery
  The time from start of treatment to the date of death from any cause or last follow-up date
Short-term surgery outcomes | 2 weeks after surgery
  Operation time, blood loss during surgery, transfusion requirement during surgery, and complication rate within 2 weeks following surgery
Safety and tolerability of nivolumab | 6 months
  The incidence, severity as graded by NCI CTCAE v5.0, seriousness and relationship to study medication of adverse events (AEs)

OTHER OUTCOMES:
Exploratory analyses | within 1 year after treatment completion of the last subject
  Exploration of potential biomarkers predicting treatment response to nivolumab using biological specimens collected

CONTACTS AND LOCATIONS:
Overall Officials: Tan-to Cheung, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- See also: HKU Clinical Trials Registry record — http://www.hkuctr.com/Study/Show/1aa3c360332c4a72abe5db565b152349